CLINICAL TRIAL: NCT01009944
Title: Genetic Mechanisms in Human Hypertension RAAS Inhibition Study
Brief Title: Genetic Mechanisms in Human Hypertension Renin-angiotensin-aldosterone System (RAAS) Inhibition Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Gordon H. Williams, MD, Chief, Cardiovascular Endocrinology Section, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007p002290
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Hypertension
Keywords: High blood pressure
MeSH Terms: conditions — Hypertension | interventions — Lisinopril; Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lisinopril, Atenolol (Experimental)
  Interventions: Drug: Lisinopril, Atenolol

INTERVENTIONS:
Drug: Lisinopril, Atenolol — once a day for 14 weeks
  Other Names: Tenormin (Atenolol); Prinivil, Zestril (Lisinopril)

SUMMARY:
The purpose of this study is to develop an approach to provide personalized medicine to individuals who have hypertension (high blood pressure). The investigators plan to use people's genetic characteristics (traits) to determine what medication they should use to lower their blood pressure most effectively. The investigators will give individuals one of two medications to treat hypertension (lisinopril or atenolol). The investigators believe that depending on the individuals genetic background one medication will work better in lowering their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female hypertensive participants who were previously studied in SCOR program.

Exclusion Criteria:

* Diabetes
* Taking other medications beside thyroid or estrogen supplements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
One type of blood pressure medication will better treat individuals with certain genetic backgrounds. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gordon H. Williams, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States